CLINICAL TRIAL: NCT00707382
Title: A Three-armed Randomised Controled Trial on the Effect of Genotyping for CYP450 Polymorphisms and Intense Clinical Monitoring on Antipsychotic Drug Treatment.
Brief Title: Effect of Genotyping for CYP450 Polymorphisms Versus Intense Clinical Monitoring on Antipsychotic Drug Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gesche Jurgens (Other)
Collaborators: Bispebjerg Hospital (Other); Research Unit, Psyciatric Centre Bispebjerg (Unknown); Research Institute of Biological Psychiatry,Psychiatric Centre Sct. Hans (Unknown); Danish Centre for Health Technology Assessment (Other); The Ministry of Health and Prevention, Denmark (Other Government); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor-Investigator, Gesche Jurgens, MD, PhD, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H-D-2007-0056
Record Dates: First submitted 2008-06-26; First posted 2008-06-30 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Schizophrenia
Keywords: Pharmacogenetics; Compliance; Antipsychotic drugs; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Patient Compliance | interventions — Genotype

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Genotyping for CYP4502D6 and 2C19 polymorphisms (Other): In this study arm (1) the genotype information is given to the physician in charge of treatment and can be used to direct the pharmacological treatment in accordance with the current guidelines from Sct. Hans hospital. In the guidelines the genotype is translated to the clinical designation "normal", "slow" or "fast" metabolizer of CYP2D6 or "normal" or "slow" metabolizer of CYP2C19. Different treatment options for the different genotypes are described in the clinical guidelines.
  Interventions: Genetic: (1) Genotyping for CYP4502D6 and 2C19 polymorphisms
- (2) Intense clinical monitoring (Other): In this study arm (2) the genotype information is not revealed. The intervention consists of an intensified clinical monitoring of treatment effect, side effects and patient perspective. Staffpersonnel is trained in the use of a clinical manual that builds on a selection of validated questions from the Scale for the Assessment of Positive Symptoms (SAPS), Side effect score (Udvalg af Kliniske Undersøgelser (UKU) and Rating of Medical Influences (ROMI). The manual has to be used at least once in a quarter (every third month), which is monitored by the study personnel. Data registered by the patients primary contact person are not used as outcome measures in the study but only as intervention tool for the optimisation of the medical antipsychotic treatment.
  Interventions: Other: (2) Intense clinical monitoring
- (3) Control (No Intervention): In this studyarm (3), (Control) treatment followed usual local practice. The genotype information was not revealed.
  Interventions: Other: (3) Control

INTERVENTIONS:
Genetic: (1) Genotyping for CYP4502D6 and 2C19 polymorphisms — In this study arm (1), the genotype information is given to the physician in charge of treatment and can be used to direct the pharmacological treatment according to local guidelines. In the guidelines the genotype is translated to the clinical designation "normal", "slow" or "fast" metabolizer of CYP2D6 or "normal" or "slow" metabolizer of CYP2C19. Different treatment options for the different genotypes are described.
  Arms: Genotyping for CYP4502D6 and 2C19 polymorphisms
Other: (2) Intense clinical monitoring — In this study arm (2) the genotype information is not revealed. The intervention consists of an intensified clinical monitoring of treatment effect, side effects and patient perspective. Staffpersonnel is trained in the use of a clinical manual that builds on a selection of validated questions from the Scale for the Assessment of Positive Symptoms (SAPS), Side effect score (Udvalg af Kliniske Undersøgelser (UKU) and Rating of Medical Influences (ROMI). The manual has to be used at least once in a quarter (every third month), which is monitored by the study personnel. Data registered by the patients primary contact person are not used as outcome measures in the study but only as intervention tool for the optimisation of the medical antipsychotic treatment.
  Arms: (2) Intense clinical monitoring
Other: (3) Control — In this studyarm (3), (Control) treatment followed usual local practice. The genotype information was not revealed.
  Arms: (3) Control

SUMMARY:
The purpose of this study is to determine whether genotyping for CYP2D6 and 2C19 polymorphisms or intense clinical monitoring of treatment and adverse effects improves the antipsychotic treatment in patients with schizophrenia. This study is designed as a three-armed prospective randomized controlled clinical trial and includes 300 patients with schizophrenia. Patients are followed for a period of one year.

During the study period the following effect measures are registered:

* Time to discontinuation of all antipsychotic medications
* Number of changes in medication dose
* Number of changes in medication
* Compliance (patients´ adherence to medical treatment)
* Clinical symptoms
* Adverse effects

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with schizophrenia
* Able to give written informed consent

Exclusion Criteria:

* Genotyped prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2008-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Time to discontinuation of initial antipsychotic treatment | one year

SECONDARY OUTCOMES:
Compliance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Gesche Jürgens, MD, phd, Principal Investigator — Department of Clinical Pharmacology, Bispebjerg University Hospital
Locations (1):
- Department of Clinical Pharmacology, Bispebjerg Hospital and Research Unit, Psychiatric Centre Bispebjerg, Copenhagen, Denmark

REFERENCES:
- [Derived] Jurgens G, Andersen SE, Rasmussen HB, Werge T, Jensen HD, Kaas-Hansen BS, Nordentoft M. Effect of Routine Cytochrome P450 2D6 and 2C19 Genotyping on Antipsychotic Drug Persistence in Patients With Schizophrenia: A Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2027909. doi: 10.1001/jamanetworkopen.2020.27909. PMID 33284338